CLINICAL TRIAL: NCT03054012
Title: Accuracy and Outcome of Computer-assisted Surgery for Bony Micro-vascular Reconstruction in the Head and Neck Region
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, head of department, AZ Sint-Jan AV
Other Study IDs: B0492017629990
Record Dates: First submitted 2017-02-13; First posted 2017-02-15 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Mandibular Injuries
Keywords: CAD-CAM software; accuracy; head and neck region; mandibular reconstruction
MeSH Terms: conditions — Mandibular Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CAS group: computer-assisted surgery group

SUMMARY:
Background:

Functional and aesthetic reconstruction of mandibular defects due to tumour invasion, osteoradio- or chemonecrosis or trauma are challenging. Surgeons aim to achieve a good anatomic and symmetric reconstruction with stable occlusion and condylar position. Classically this was obtained by (pre)bending a reconstruction plate, and providing osteotomies at the vascularized free flap. Today there is the availability of CAD-CAM software enabling a preoperative planning based on 3D models. This computer-assisted surgery (CAS) procedure is said to improve accuracy of the postoperative result, as well as a reduce ischemia time. However, there is a need for objective analysis of the accuracy of CAS, as well as the effective reduction in operating time and financial implication.

Study design:

Retrospective study.

All patients undergoing bony reconstruction by free vascularised flap between January 2013 and August 2016 will be included. Accuracy will be measured between the planned and actual result, through segmentation of the mandible in Brainlab software. Parameters regarding ischemic time and financial cost will be obtained from the medical files.

ELIGIBILITY:
Inclusion Criteria:

* patients of all ages
* patients of both genders
* patients requiring mandibular reconstruction due to tumour invasion, osteoradionecrosis, osteochemonecrosis or trauma
* all patients undergoing bony reconstruction by free vascularised flap
* all patients treated between January 2013 and August 2016
* all patients where CAS was applied

Exclusion Criteria:

* all patients not eligible according to abovementioned criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients undergoing bony reconstruction by free vascularised flap between January 2013 and August 2016 will be included
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
accuracy of planned and actual result, through segmentation of mandibles Brainlab software | 6 months postoperative

SECONDARY OUTCOMES:
ischemia time | perioperative
financial implication | preoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — Head of department

IPD SHARING:
Plan to Share IPD: No